CLINICAL TRIAL: NCT03830645
Title: Platelet Rich Plasma in Secondary Spontaneous Pneumothorax
Brief Title: PRP in 2ry Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmad Abbas, Principal investigator &lecturer of chest disases zagazig university, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#4931-4-11-2018
Record Dates: First submitted 2019-01-27; First posted 2019-02-05 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Pneumothorax Spontaneous Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet rich plasma group (Experimental)
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Application of platelet rich plasma through the intercostal tube into the pleural space

SUMMARY:
secondary spontaneous pneumothorax patients will be enrolled ,all of them will receive PRP with different doses and schedules

ELIGIBILITY:
Inclusion Criteria:

* COPD patients developed spontanous pneumothorax and was managed with intercostal tube insertion

Exclusion Criteria:

* refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Air leak assessment by Cerfolio classification of the air leak by single observer | within 10 days after application of platelet rich plasma
  Continuous:Air leak is Present throughout the respiratory cycle Inspiratory : Present during the inspiration phase of the respiratory cycle. Expiratory: Present only during the expiratory phase of the respiratory cycle Forced expiration: Present only when the patient coughs or forces exhalation
physician assessment of complete lung inflation by absence of signs of pneumothorax in chest x ray done to the patient during hospital stay | within 10 days after application of platelet rich plasma
  no Chest x ray signs of pneumothorax i.e no jet balck translucency or border of collapsed lung) by physician interpretation
recurrence of pneumothorax by physician interpretation of Chest x ray done to the patient in follow up visit i.e detecting jet balck translucency or border of collapsed lung | one month after removal of intercostal tube
  no Chest x ray signs of pneumothorax i.e no jet balck translucency or border of collapsed lung) by physician interpretation
recurrence of pneumothorax by physician interpretation of Chest x ray done to the patient in follow up visit i.e detecting jet balck translucency or border of collapsed lung | two months after removal of intercostal tube
  no Chest x ray signs of pneumothorax i.e no jet balck translucency or border of collapsed lung) by physician interpretation
recurrence of pneumothorax by physician interpretation of Chest x ray done to the patient in follow up visit i.e detecting jet balck translucency or border of collapsed lung | three months after removal of intercostal tube
  no Chest x ray signs of pneumothorax i.e no jet balck translucency or border of collapsed lung) by physician interpretation
recurrence of pneumothorax by physician interpretation of Chest x ray done to the patient in follow up visit i.e detecting jet balck translucency or border of collapsed lung | six months after removal of intercostal tube
  no Chest x ray signs of pneumothorax i.e no jet balck translucency or border of collapsed lung) by physician interpretation

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of medicine Chest Department, Zagazig, Asharqia, Egypt